CLINICAL TRIAL: NCT00382304
Title: A Study of the Pharmacokinetics of GT267-004 in Patients With Clostridium Difficile-Associated Diarrhea
Brief Title: A Study of the Absorption of GT267-004 in Patients With Clostridium Difficile-Associated Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOL26700606
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Pseudomembranous Colitis; Clostridium Difficile Diarrhea; Antibiotic-Associated Diarrhea
Keywords: Clostridium difficile-associated diarrhea; C. difficile; CDAD; Clostridium difficile; Clostridium difficile Disease; Clostridium Enterocolitis; Antibiotic-Associated Colitis; Infectious diarrhea
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Dysentery

INTERVENTIONS:
Drug: tolevamer potassium-sodium (GT267-004)

SUMMARY:
Approximately 24 patients will be entered into this study taking place in Canada. The aim of this study is to determine if an investigational drug is absorbed (taken up) in patients with C. difficile-associated diarrhea (CDAD). The investigational drug will be given in addition to current standard antibiotic treatment so that all patients will receive active medication. All study related care is provided including doctor visits, physical exams, laboratory tests, and study medication. The total length of participation is approximately 7 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* The presence of CDAD at the time of enrollment with no other likely etiology for the diarrhea

Exclusion Criteria:

* > 72 hours of treatment with metronidazole, vancomycin, or other antibacterial therapy specifically targeting the current acute episode of CDAD
* Patient not considered sufficiently stable clinically to complete the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The extent of GT267-004 absorption as measured in the blood and urine by pharmacokinetic analysis

SECONDARY OUTCOMES:
Safety as measured by physical examinations (including vital signs), adverse events and changes in safety laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- Canada (8):
  - Edmonton, Alberta
  - Nanaimo, British Columbia
  - Vancouver, British Columbia
  - Ottowa, Ontario
  - Richmond Hill, Ontario
  - Montreal, Quebec
  - Rimouski, Quebec
  - Sherbrooke, Quebec